CLINICAL TRIAL: NCT00673595
Title: Endothelial Function and Autonomic Regulation After Short-term Smoking Cessation: Varenicline Versus Placebo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruiting sujects and subjects complying with the protocol
Sponsor: Mayo Clinic (Other)
Responsible Party: John H. Eisenach, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 06-007194
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-02

CONDITIONS: Smoking
Keywords: smoking; varenicline; flow-mediated dilation; blood pressure; baroreflex
MeSH Terms: conditions — Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Active Comparator): Participants on this arm will receive varenicline tablets for 15 days.
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): Participants on this arm will receive placebo tablets for 15 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Smoking cessation assistance: study days 1-3: 0.5 mg once daily, study days 4-7: 0.5 mg twice daily, study days 8-15: 1 mg twice daily; study day 16: 1 mg once. The tablets should be taken orally after food intake with 200 ml of water.
  The treatment phase may be prolonged up to a maximum of 2 weeks under the following conditions: 1) the participant voluntarily agrees to the prolongation of the study, 2) both the participant and investigator are confident that the participant will be able to completely refrain from smoking for at least 10 days until the final study day.
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — The pharmacy will prepare tablets that match the varenicline tablets. The tablets should be taken orally after food intake with 200 ml of water.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate endothelial function and autonomic regulation (for example, heart rate and blood pressure) in smokers before and after short-term smoking cessation. The endothelium is the thin layer of cells that lines the interior surface of blood vessels. The endothelium releases nitric oxide, which promotes dilation of the blood vessels and inhibits inflammation. Previous studies have shown that tobacco use is associated with endothelial dysfunction, and tobacco use increases heart rate and blood pressure.

We hypothesize that 2 weeks of smoking cessation will improve endothelial function. We will also determine if endothelial function and autonomic regulation after short-term smoking cessation differs for patients that achieve abstinence with the smoking cessation agent varenicline compared to placebo.

DETAILED DESCRIPTION:
Smoking is a major cardiovascular risk factor and is associated with arterial endothelial dysfunction, a key event in atherosclerosis. Previous observations have suggested that smoking-related endothelial dysfunction is dose-related and potentially reversible after withdrawal from smoking. To our knowledge, no data are available regarding potential improvement of arterial endothelial function in the first weeks of smoking cessation. This time frame is especially important because due to smoke-free policies in healthcare facilities, all smokers requiring surgery are abstinent from tobacco for at least some period of time.

Varenicline, a partial agonist at α4β2 neuronal nicotinic acetyl-choline (nAChR) receptors, received FDA approval as a novel medication for helping cigarette smokers to stop smoking. Given the anticipated common use of varenicline, it is important to define if the drug alters endothelial function and/or autonomic effects. Based on the lesser potency of varenicline (compared to nicotine) at nAChR receptors in peripheral ganglia and on endothelial cells of blood vessels, it may be hypothesized that varenicline has less or no influence on autonomic control of blood pressure and heart rate, and less or no influence on endothelial function.

Therefore, the aims of this study are 1) to determine the effects of short-term smoking cessation on endothelial function and autonomic regulation, and 2) to determine if these effects will be altered during treatment with varenicline.

ELIGIBILITY:
Inclusion Criteria:

* Regular smokers (currently >10 cigarettes/day; >5 pack years)
* Willing to quit smoking for at least the duration of the study
* Able and willing to give written informed consent

Exclusion Criteria:

* Known condition causing endothelial dysfunction except smoking (i.e. diabetes, hyperlipi¬demia, arterial hypertension, obesity)
* Regular drug treatment and/or sporadic consumption of drugs within the last 4 weeks (exclusion has to be decided in each individual)
* Acute or chronic illness
* Participation in clinical trial within 1 month before the study
* Excessive daily intake of alcohol (>2 servings per day) or caffeine (>4 servings/day)
* Drug and/or alcohol abuse.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2007-03; Primary Completion 2009-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Eisenach, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Mayo Clinic in Rochester, Minnesota from March 2007 to February 2009.
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 8 | 11
Completed | 8 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 11 | 19
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Arterial Endothelial Function as Measured by Flow-mediated Dilation
Description: Flow-mediated dilation of the brachial artery will be measured using high-resolution ultrasound. Arterial diameter will be measured above the small cavity in the elbow joint from ultrasound images at rest in response to an increase in blood flow to the area. This blood flow will be induced by inflation of a blood pressure cuff placed around the forearm to a pressure of at least 50 mm Hg above systolic pressure for 5 min, followed by release. The ultrasound image of the artery will be recorded continuously from 30 sec before until 2 min after cuff release.
Time Frame: 2 weeks after participants quit smoking (study visit 3, day 15)
Population: This study was terminated early due to difficulty with recruiting subjects and with subjects complying with the protocol; analysis was not performed.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: 24-hour Ambulatory Blood Pressure
Description: Ambulatory blood pressure will be measured using the Spacelabs 90202 recorder. Systolic and diastolic blood pressure during the 24-hour period will be analyzed.
Time Frame: 2 weeks after participants quit smoking (study visit 3, day 15)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events from randomization through 2 weeks after participants quit smoking (study visit 3, day 15).
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/8 | 0/11

LIMITATIONS AND CAVEATS:
This study was terminated early due to difficulty with recruiting subjects and with subjects complying with the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes